CLINICAL TRIAL: NCT01255735
Title: Randomized Controlled Trial of Voice on Children With Vocal Nodules
Status: Completed | Type: Observational
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: Drexel University College of Medicine (Other); Medical College of Wisconsin (Other); The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Other Study IDs: 10-04-024
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-11

CONDITIONS: Vocal Fold Nodules
Keywords: pediatrics; voice; voice therapy; vocal therapy; hoarseness
MeSH Terms: conditions — Hoarseness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Vocal nodules: Two groups of children who are hoarse and have vocal nodules will be examined to see whether voice therapy is effective as a treatment strategy

SUMMARY:
The primary objective of this study is to determine the impact of voice therapy on voice-related quality of life in children age 6-10 years old with apparent vocal fold nodules, as measured by the validated Pediatric Voice-Related Quality of Life Instrument (PVRQOL)administered 4 weeks after completion of voice therapy.

DETAILED DESCRIPTION:
Voice disorders place over five million school-aged children at increased risk for inferior school performance, dysfunctional social development, and higher participation in criminal activities. The lesions most commonly associated with pediatric vocal dysfunction are reported to be vocal fold nodules, which are present in up to 21% of the general pediatric population and are associated with behavioral problems and inferior quality of life. Voice therapy with a speech-language pathologist is recommended by 95% of otolaryngologists for management of vocal fold nodules. When implemented, this voice therapy requires significant time investment and typically results in regular absence from the classroom over a period of 1-3 months or longer, depending on the protocol and the setting. Regular absence from school has been shown to place children at risk for poorer scholastic performance but the benefits of this voice therapy have yet to be demonstrated in any rigorous prospective, controlled trial. Thus, the most widely used treatment for the most common lesion associated with pediatric voice disorders has not been rigorously tested in a randomized controlled trial to determine whether it may have benefits.

A randomized clinical trial addressing whether voice therapy improves voice-related quality of life for children with apparent vocal fold nodules is a logical step toward developing an evidence-based treatment plan to optimize outcomes for this sizable population of at-risk children. There are currently no well-powered, prospective, controlled studies which compare voice therapy versus control in children who present with apparent nodules. Our goal is to remedy this deficiency through testing of the following primary null hypothesis: There is no difference in the change in PVRQOL scores after 3 months of treatment with voice therapy versus office instructions.

ELIGIBILITY:
Inclusion criteria

1. Eligibility is contingent on the presence of apparent vocal fold nodules, which are defined as bilateral, localized, benign, superficial growths with protrusion on the medial surface of the true vocal folds at the junction of their anterior and middle thirds. This examination is based on video-stroboscopic examination, or, in rare cases, on operative microsuspension laryngoscopy. In addition, strict exclusion criteria are applied toward excluding masses that are not nodules. Defining characteristics for these inclusion criteria are based upon the evaluations of three senior otolaryngologists of each participant's exam. Children evaluated by the senior otolaryngologist at each institution suspected to have vocal fold nodules are candidates for inclusion to this study. Patient de-identified images of the stroboscopy are reviewed by each of the other two laryngologists; only those children with confirmed vocal fold nodules by the all three senior otolaryngologists will be considered for entry into this study.
2. Children 6 to10 years of age will be enrolled. The rationale for this age range was previously noted. In brief, children in this age range (a) have similar educational and social exposures; (b) will likely not yet encounter pubertal changes affecting the larynx; and (c) are relatively cognitively homogeneous. Moreover, children in this age range have the ability to cooperate with voice therapy and have also been shown to be tolerant of stroboscopic examination. Finally, the voice therapy regimen in this protocol has been shown to be clinically effective for many children in this age range.
3. Voice-related quality of life must be affected to the extent that baseline PVRQOL scores are <87.5 (on a scale of the worst, 0, to the best, 100) at the time of entry into the trial. Based on previously published data, this subset of scores will be clearly distinct from scores in children with normal voices. In addition, scores <87.5 represent worse than average scores among children diagnosed with vocal fold nodules.
4. Dysphonia duration prior to randomization must be at least 12 weeks, in order to ensure that vocal dysfunction is chronic in nature.
5. Hearing in better ear of 35 dB or better.
6. Agreement by informed consent from the parents and informed assent from the child participant with anticipated commitment to compliance throughout the follow up period of 3 months is necessary for enrollment which includes time commitment of up to 3 hours per week to therapy sessions and homework.
7. Vocal fold nodules are a pathology that predominantly affects males. A number of studies and the databases utilized to track this pathology at the clinical sites indicate that the male: female ratio is approximately 7:3. Given this background, the enrollment plan for the current investigation will seek to have a 30% female representation of the patients enrolled in this study to ensure appropriate gender representation. Additionally, patients with a diagnosis of pediatric vocal fold nodules predominantly are found in Caucasian populations. However, in accordance with the National Institute of Health Revitalization Act of 1993 the inclusion of minorities in this proposal will be targeted to the representation of minorities in the greater Boston, Philadelphia and Milwaukee metropolitan regions.

Exclusion criteria

1. Children with non-standard nodules or masses that are not unequivocally nodules are excluded, including those with irregular epithelium, concern for malignancy requiring biopsy, rapid growth pattern, airway obstruction requiring urgent or operative intervention, and prior laryngeal surgery. Furthermore, since there are several lesions that can present as bilateral true vocal fold masses (such as unilateral cysts or polyps with contralateral fibrovascular reaction, contact granulomas, and Reinke's edema), masses with the following characteristics will be excluded: a) yellow or blue color suggestive of a mucous- or fluid-filled component, b) pink friable lesions at the posterior aspect of the true vocal folds, c) watery edematous expansion without a distinct protrusive mass. Defining characteristics for these exclusion criteria are determined and corroborated by the evaluations of three senior otolaryngologists of each participant's videostroboscopic exam. This examination is based on video-stroboscopy, or, in rare cases, on operative microsuspension laryngoscopy. The video images will be placed on a password-protected server to which all three senior investigators will have access; these video images will not contain any patient identifying information but rather a study number that will be assigned to each participant. In addition, strict inclusion criteria are applied toward excluding masses that are not nodules.
2. Children who have previously received any form of speech therapy targeting voice and/or resonance with the exception of articulation or speech therapy.
3. Children for whom voice therapy protocols will be problematic are excluded: developmental delay, cognitive disorder, behavioral disorder, neurologic disorder, articulation disorder, phonological disorder, language disorder, expressive and/or receptive language delay, specific language impairment, central auditory processing disorder, fluency disorder, prior knowledge of voice therapy principles through previous interventions (with the exception of articulation or speech therapy), and inability to commit to at least 12 weeks of therapy as determined and evaluated by the treating speech language pathologist and confirmed by consensus of all three PIs.
4. Children whose caregivers cannot complete the primary endpoint are excluded: non-English speaking as the PVRQOL instrument is administered in English, and those unable to commit to the 3-month treatment and follow-up schedule.
5. Children whose caregivers are not willing to commit up to 3 hours per week to vocal therapy including therapy sessions and homework for up to 12 weeks.
6. Children who cannot tolerate a conscious video-stroboscopic examination and whose parents feel that the diagnostic information gained by a planned examination under anesthesia is not valuable for the severity of presenting symptoms are excluded.
7. Children with significant confounders of voice-related quality of life are excluded: vocal fold paralysis, neurologic disorder of the larynx (dystonias, tics, tremors, etc), ongoing acute upper respiratory tract infection (defined by at least 2 of the following: sneezing, coughing, nasal congestion, runny nose, or temperature greater than 100.4° F (38.0° C), and untreated or unsuccessfully treated allergic rhinitis/post nasal drip.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children ages 6-10 who have hoarseness and vocal nodules
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2011-01; Primary Completion 2015-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Pediatric Voice-Related Quality of Life Instrument (PVRQOL) | Administered at Screening, Baseline, Therapy Completion, and Follow-Up
  The PVRQOL consists of 10 questions completed by parent proxy administration that requires approximately 5 minutes to complete. It measures the parent's assessment of their child's overall quality of life as related to their vocal condition.

SECONDARY OUTCOMES:
"Consensus Auditory-Perceptual Evaluation of Voice" (CAPE-V) | Completed at Baseline, Therapy Completion, and Follow-Up
  The CAPE-V specifies standardized procedures for the perceptual evaluation of voice, including standardized recording conditions, word stimuli and rating procedures.
Phonation Threshold Pressure (PTP) | Completed at Baseline, Therapy Completion, and Follow-Up
  The aerodynamic measures obtained will focus on estimated Phonation Threshold Pressure (PTP), defined as the minimum amount of subglottal pressure required to initiate and sustain vocal fold oscillation. These measures will be obtained in a non-invasive manner from oral pressures generated during repetitive production of five consonant-vowel-consonant (CVC) strings (/pae pae pae pae pae/.
Harmonics-to-Noise Ration [HNR) | Completed at Baseline, Therapy Completion, and Follow-Up
  Recordings will be analyzed using KayPENTAX's Computerized Speech Lab (CSL). To analyze the steady state vowel productions, the steadiest one second segment from the mid portion of each vowel production will be selected from the digitized waveform for analysis, and HNR results for that segment will be obtained using CSL software.
Nodule grade | Completed at Baseline and Follow-Up
  A grading system for vocal fold nodules has been validated with established inter-rater reliability for nodule presence and size. The 3-point grading scale for nodule size will be used with grade 1 being small, grade 2 a moderate nodule, and grade 3 a large nodule. The contour of the nodule will also be rated as either discrete or sessile. One secondary objective of the study is to compare nodule grade across baseline and 12 (or 16) weeks. Changes in grade are compared for subjects treated with voice therapy versus office instructions alone.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hartnick, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (4):
- United States (3):
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Drexell University College of Medicine, Philadelphia, Pennsylvania
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- The Hospital For Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Hartnick C, Ballif C, De Guzman V, Sataloff R, Campisi P, Kerschner J, Shembel A, Reda D, Shi H, Sheryka Zacny E, Bunting G. Indirect vs Direct Voice Therapy for Children With Vocal Nodules: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2018 Feb 1;144(2):156-163. doi: 10.1001/jamaoto.2017.2618. PMID 29270612